CLINICAL TRIAL: NCT03868111
Title: Comparison Between Sufentanil and Remifentanil as General Anesthetic Adjuvant
Brief Title: Sufentanil as Adjuvant of Balanced Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoung-Ho Ryu, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-02-001
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil (Experimental): Balanced anesthesia is maintained with 1 MAC desflurane and sufentanil during laparoscopic cholecystectomy.
  Interventions: Drug: Sufentanil
- Remifentanil (Experimental): Balanced anesthesia is maintained with 1 MAC desflurane and remifentanil during laparoscopic cholecystectomy.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Sufentanil — The infusion rate of sufentanil is adjusted to achieve a surgical pleth index of 20-50 throughout the operative time.
  Other Names: Group S
  Arms: Sufentanil
Drug: Remifentanil — The infusion rate of remifentanil is adjusted to achieve a surgical pleth index of 20-50 throughout the operative time.
  Other Names: Group R
  Arms: Remifentanil

SUMMARY:
The aim of the study was to compare the efficacy and safety between sufentanil and remifentanil as an adjuvant of balanced general anesthesia.

DETAILED DESCRIPTION:
The investigators hypothesized that sufentanil would reduce postoperative pain than remifentanil without prolonging recovery times in minor laparoscopic surgery when administered equivalent antinociceptive doses during surgery. Intraoperative opioid administration for equivalent nociception-antinociception balance could be achieved via surgical pleth index (SPI)-guided analgesia. This study was designed to compare the efficacy and safety between sufentanil and remifentanil as an adjuvant of balanced anesthesia in patients undergoing laparoscopic cholecystectomy under SPI-guided opioid administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 19 and 65 years
* Patients with American Society of Anesthesiologists physical status I or II
* Patients scheduled for elective laparoscopic cholecystectomy under balanced general anesthesia for benign cholecystic diseases
* Patients obtaining written informed consent

Exclusion Criteria:

* Patients with asthma or hypertension
* Patients with an inability to express their pain accurately
* Patients with an inability to understand the pain scale
* Patients with chronic abdominal pain or chronic pain syndrome
* Patients who required to convert to laparotomy from laparoscopic surgery
* Patients who required to receive incidental lower abdominal procedures owing to adhesion, injury, or other incidental findings at the lower abdominal cavity
* Patients with a history of drug or alcohol abuse
* Pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Postoperative wound pain score | 10 minutes after surgery
  The pain score is evaluated by 10 point visual analogue scale at post-anesthesia care unit. The visual analogue scale is presented as a 10-cm line with verbal descriptors indicating "no pain" and "pain as bad as it could be". The visual analogue scale ranges from 0 to 10, representing minimum and maximum pain levels, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Ho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea